CLINICAL TRIAL: NCT06601855
Title: Cholecystectomy Could be Performed in Adults Older Than 80 Years Old With Mild to Moderate Acute Cholecystitis
Brief Title: Cholecystectomy Could be Performed in Older Adults With Acute Cholecystitis
Status: Completed | Type: Observational
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: jessie21211
Record Dates: First submitted 2024-09-15; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Acute Cholecystitis
Keywords: acute cholecystitis; aged; cholecystectomy
MeSH Terms: conditions — Cholecystitis, Acute | interventions — Cholecystectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cholecystectomy group: Patient in this group received cholecystectomy, whether immediately, or delayed
  Interventions: Procedure: Cholecystectomy
- Non-operative management group: Patients in this group did not receive cholecystectomy during follow up period

INTERVENTIONS:
Procedure: Cholecystectomy — Cholecystectomy, whether open or laparoscopic
  Groups: Cholecystectomy group

SUMMARY:
The goal of this retrospective cohort observational study is to learn about the long-term and short-term effects of cholecystectomy in people aged 80 or over the age of 80, who have mild to moderate acute cholecystitis. The main question it aims to answer is:

Does cholecystectomy bring harm or benefit to people aged 80, or over the age of 80, who have mild to moderate acute cholecystitis? People who received cholecystectomy are compared to those who did not, for short- and long-term outcomes, with a follow up period for 18 months.

DETAILED DESCRIPTION:
All data were collected from Shuang-Ho Hospital electronic medical record.

ELIGIBILITY:
Inclusion Criteria:

* Acute cholecystitis patients aged 80 years or older

Exclusion Criteria:

* Grade III acute cholecystitis
* Concurrent cholangitis, common bile duct stones, pancreatitis, gallbladder cancer, hepatocellular carcinoma, periampullary cancer
* Received other operations at the same admission other than cholecystectomy
* Discharged against advice of physician
* Received further management at another hospital for acute cholecystitis

Min Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients with mild to moderate (grade I and grade II) acute cholecystitis, who were 80 years old or older, were included.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | From admission to discharge, average 8 days, minimal 2 days, maximal 51 days
  Expired during admission
30-day mortality | 30 days since discharge
  Expired within 30 days since discharge
Hospital return rate | 18 months after discharge
  Rate of return to emergency room or readmission after discharge

SECONDARY OUTCOMES:
Hospital length of stay | From admission to discharge, average 8 days, minimal 2 days, maximal 51 days
  Period of hospitalization
Intensive care unit length of stay | From admission to discharge, average 8 days, minimal 2 days, maximal 51 days
  How long has the person been admitted to the intensive care unit
Intensive care unit admission frequency | From admission to discharge, average 8 days, minimal 2 days, maximal 51 days
  How many times have the person been admitted to the intensive care unit
Outpatient department follow up frequency | 18 months after discharge
  How many times has the person visited the outpatient department since discharge due to gallstone related disease or post cholecystectomy
Outpatient department follow up duration | 18 months after discharge
  Period of the last visit to the outpatient department due to gallstone related disease or post cholecystectomy, since discharge

CONTACTS AND LOCATIONS:
Overall Officials: Chieh-Ju Liao, MD, Principal Investigator — Taipei Medical University-Shuang Ho Hospital,Ministry of Health and Welfare; Kuei-Yen Tsai, PhD, Principal Investigator — Taipei Medical University-Shuang Ho Hospital,Ministry of Health and Welfare
Locations (1):
- Taipei Medical University-Shuang Ho Hospital,Ministry of Health and Welfare, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Escartin A, Gonzalez M, Cuello E, Pinillos A, Muriel P, Merichal M, Palacios V, Escoll J, Gas C, Olsina JJ. Acute Cholecystitis in Very Elderly Patients: Disease Management, Outcomes, and Risk Factors for Complications. Surg Res Pract. 2019 Feb 3;2019:9709242. doi: 10.1155/2019/9709242. eCollection 2019. PMID 30854417
- [Background] Asbun, Horacio & Shah, Mihir & Ceppa, Eugene & Auyang, Edward. (2020). The SAGES Manual of Biliary Surgery. 10.1007/978-3-030-13276-7
- [Background] Yetkin G, Uludag M, Oba S, Citgez B, Paksoy I. Laparoscopic cholecystectomy in elderly patients. JSLS. 2009 Oct-Dec;13(4):587-91. doi: 10.4293/108680809X1258998404604. PMID 20202402
- [Background] Lee SJ, Choi IS, Moon JI, Yoon DS, Lee SE, Sung NS, Kwon SU, Bae IE, Roh SJ, Choi WJ. Elective Laparoscopic Cholecystectomy Is Better than Conservative Treatment in Elderly Patients with Acute Cholecystitis After Percutaneous Transhepatic Gallbladder Drainage. J Gastrointest Surg. 2021 Dec;25(12):3170-3177. doi: 10.1007/s11605-021-05067-1. Epub 2021 Jun 25. PMID 34173163
- [Result] Pisano M, Allievi N, Gurusamy K, Borzellino G, Cimbanassi S, Boerna D, Coccolini F, Tufo A, Di Martino M, Leung J, Sartelli M, Ceresoli M, Maier RV, Poiasina E, De Angelis N, Magnone S, Fugazzola P, Paolillo C, Coimbra R, Di Saverio S, De Simone B, Weber DG, Sakakushev BE, Lucianetti A, Kirkpatrick AW, Fraga GP, Wani I, Biffl WL, Chiara O, Abu-Zidan F, Moore EE, Leppaniemi A, Kluger Y, Catena F, Ansaloni L. 2020 World Society of Emergency Surgery updated guidelines for the diagnosis and treatment of acute calculus cholecystitis. World J Emerg Surg. 2020 Nov 5;15(1):61. doi: 10.1186/s13017-020-00336-x. PMID 33153472
- [Result] Wiggins T, Markar SR, Mackenzie H, Jamel S, Askari A, Faiz O, Karamanakos S, Hanna GB. Evolution in the management of acute cholecystitis in the elderly: population-based cohort study. Surg Endosc. 2018 Oct;32(10):4078-4086. doi: 10.1007/s00464-018-6092-5. Epub 2018 Jul 25. PMID 30046948
- [Result] Lee CE, Lee SJ, Moon JI, Choi IS, Yoon DS, Choi WJ, Lee SE, Sung NS, Kwon SU, Bae IE, Roh SJ, Kim SG. Acute cholecystitis in old adults: the impact of advanced age on the clinical characteristics of the disease and on the surgical outcomes of laparoscopic cholecystectomy. BMC Gastroenterol. 2023 Sep 25;23(1):328. doi: 10.1186/s12876-023-02954-6. PMID 37749524
- [Result] Loozen CS, van Santvoort HC, van Duijvendijk P, Besselink MG, Gouma DJ, Nieuwenhuijzen GA, Kelder JC, Donkervoort SC, van Geloven AA, Kruyt PM, Roos D, Kortram K, Kornmann VN, Pronk A, van der Peet DL, Crolla RM, van Ramshorst B, Bollen TL, Boerma D. Laparoscopic cholecystectomy versus percutaneous catheter drainage for acute cholecystitis in high risk patients (CHOCOLATE): multicentre randomised clinical trial. BMJ. 2018 Oct 8;363:k3965. doi: 10.1136/bmj.k3965. PMID 30297544
- [Result] Ramirez-Giraldo C, Venegas-Sanabria LC, Rojas-Lopez S, Avendano-Morales V. Outcomes after laparoscopic cholecystectomy in patients older than 80 years: two-years follow-up. BMC Surg. 2024 Mar 12;24(1):87. doi: 10.1186/s12893-024-02383-6. PMID 38475792